CLINICAL TRIAL: NCT02633488
Title: Effect of Metformin on Insulin Sensitivity and Pan-Arterial Vascular Function in Adults With Metabolic Syndrome
Acronym: EJB044
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Eugene Barrett, MD PhD, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16121
Record Dates: First submitted 2014-09-26; First posted 2015-12-17 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome; Insulin Sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 12 weeks of Placebo tablet 3 x daily
  Interventions: Drug: Placebos
- Metformin (Experimental): 12 weeks of Metformin tablet 850 mg 3 x daily
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: Placebos — A 12 week single blind placebos
  Other Names: inactive substance
  Arms: Placebo
Drug: metformin — A 12 week single blind metformin
  Other Names: glucophage
  Arms: Metformin

SUMMARY:
The purpose of this study is to look at how insulin (a hormone that helps the cells get energy from sugar) in our body affects blood vessels (elasticity in the bigger blood vessels and blood flow in the smaller blood vessels in the arm) and how Metformin (a drug that makes you more sensitive to insulin) affects insulin's action on the blood vessels.

DETAILED DESCRIPTION:
In our protocol, we will study vascular function using pulse wave velocity (PWV) augmentation index (AI), flow mediated dilation (FMD) and contrast enhanced ultrasound (CEU) as well as insulin sensitivity (euglycemic clamp) in 50 adults with metabolic syndrome, age 18-60 years. They will each be studied 4 times,before and after two 12-wk interventions (randomly assigned) as follows: 1) Placebos and 2) Metformin . This is a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60

  * No smoking the past 6 months
  * Normal screening labs or no clinically significant values-except those listed below
  * Must have 3 of the following 4 characteristics established by NCEP-AHA-NHLBI

    * Males waist circumference greater than 40 inches, females greater than 35 inches
    * Blood pressure greater than 130/85 or on treatment with one or more antihypertensive agent
    * Fasting plasma triglycerides >150 or HDL <40 (males) <50 (females)
    * Fasting blood sugar >100 but <126
  * Subject may participate if on the following drugs, provided the drugs can remain at stable doses throughout the 12 week treatment interval.

    * Ace inhibitor
    * ARB
    * HMG CoA reductase inhibitor
    * Beta blocker
    * Calcium channel blockers
    * Alpha-adrenergic antagonist

Exclusion Criteria:

* Smoking presently or in the past 6 months
* HbA1c ≥ 6.5
* Glucocorticoids-eg: prednisone, dexamethasone
* Any known sensitivity or intolerance to Metformin
* Any chronic GI disorders such as Irritable Bowel Syndrome or Crohns disease
* History of congestive heart failure, ischemic heart disease, severe pulmonary disease, liver or kidney disease.
* History of malignant or metabolic disorders including diabetes
* Presence of an intracardiac or intrapulmonary shunt (we will screen for this by auscultation during the physical exam by PI)
* Hypersensitivity to perflutren (contained in Definity)
* Pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Barett, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reported as composite for the entire population. In some figures individual data point are displayed but not identified with individual subjects.

REFERENCES:
- [Background] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Background] Brown A, Reynolds LR, Bruemmer D. Intensive glycemic control and cardiovascular disease: an update. Nat Rev Cardiol. 2010 Jul;7(7):369-75. doi: 10.1038/nrcardio.2010.35. Epub 2010 Apr 20. PMID 20404853
- [Background] Cooper-DeHoff RM, Gong Y, Handberg EM, Bavry AA, Denardo SJ, Bakris GL, Pepine CJ. Tight blood pressure control and cardiovascular outcomes among hypertensive patients with diabetes and coronary artery disease. JAMA. 2010 Jul 7;304(1):61-8. doi: 10.1001/jama.2010.884. PMID 20606150
- [Background] Steinberg HO, Paradisi G, Hook G, Crowder K, Cronin J, Baron AD. Free fatty acid elevation impairs insulin-mediated vasodilation and nitric oxide production. Diabetes. 2000 Jul;49(7):1231-8. doi: 10.2337/diabetes.49.7.1231. PMID 10909983
- [Background] Steinberg HO, Tarshoby M, Monestel R, Hook G, Cronin J, Johnson A, Bayazeed B, Baron AD. Elevated circulating free fatty acid levels impair endothelium-dependent vasodilation. J Clin Invest. 1997 Sep 1;100(5):1230-9. doi: 10.1172/JCI119636. PMID 9276741
- [Background] Tripathy D, Mohanty P, Dhindsa S, Syed T, Ghanim H, Aljada A, Dandona P. Elevation of free fatty acids induces inflammation and impairs vascular reactivity in healthy subjects. Diabetes. 2003 Dec;52(12):2882-7. doi: 10.2337/diabetes.52.12.2882. PMID 14633847
- [Background] de Jongh RT, Serne EH, Ijzerman RG, de Vries G, Stehouwer CD. Free fatty acid levels modulate microvascular function: relevance for obesity-associated insulin resistance, hypertension, and microangiopathy. Diabetes. 2004 Nov;53(11):2873-82. doi: 10.2337/diabetes.53.11.2873. PMID 15504968
- [Background] Liu Z, Liu J, Jahn LA, Fowler DE, Barrett EJ. Infusing lipid raises plasma free fatty acids and induces insulin resistance in muscle microvasculature. J Clin Endocrinol Metab. 2009 Sep;94(9):3543-9. doi: 10.1210/jc.2009-0027. Epub 2009 Jun 30. PMID 19567533
- [Background] Westerbacka J, Seppala-Lindroos A, Yki-Jarvinen H. Resistance to acute insulin induced decreases in large artery stiffness accompanies the insulin resistance syndrome. J Clin Endocrinol Metab. 2001 Nov;86(11):5262-8. doi: 10.1210/jcem.86.11.8047. PMID 11701689
- [Background] Westerbacka J, Vehkavaara S, Bergholm R, Wilkinson I, Cockcroft J, Yki-Jarvinen H. Marked resistance of the ability of insulin to decrease arterial stiffness characterizes human obesity. Diabetes. 1999 Apr;48(4):821-7. doi: 10.2337/diabetes.48.4.821. PMID 10102699
- [Background] Baron AD, Steinberg HO, Chaker H, Leaming R, Johnson A, Brechtel G. Insulin-mediated skeletal muscle vasodilation contributes to both insulin sensitivity and responsiveness in lean humans. J Clin Invest. 1995 Aug;96(2):786-92. doi: 10.1172/JCI118124. PMID 7635973
- [Background] Barrett EJ, Eggleston EM, Inyard AC, Wang H, Li G, Chai W, Liu Z. The vascular actions of insulin control its delivery to muscle and regulate the rate-limiting step in skeletal muscle insulin action. Diabetologia. 2009 May;52(5):752-64. doi: 10.1007/s00125-009-1313-z. Epub 2009 Mar 13. PMID 19283361
- [Background] Steinberg HO, Chaker H, Leaming R, Johnson A, Brechtel G, Baron AD. Obesity/insulin resistance is associated with endothelial dysfunction. Implications for the syndrome of insulin resistance. J Clin Invest. 1996 Jun 1;97(11):2601-10. doi: 10.1172/JCI118709. PMID 8647954
- [Background] Rossi R, Cioni E, Nuzzo A, Origliani G, Modena MG. Endothelial-dependent vasodilation and incidence of type 2 diabetes in a population of healthy postmenopausal women. Diabetes Care. 2005 Mar;28(3):702-7. doi: 10.2337/diacare.28.3.702. PMID 15735211
- [Background] Goldfine AB, Beckman JA, Betensky RA, Devlin H, Hurley S, Varo N, Schonbeck U, Patti ME, Creager MA. Family history of diabetes is a major determinant of endothelial function. J Am Coll Cardiol. 2006 Jun 20;47(12):2456-61. doi: 10.1016/j.jacc.2006.02.045. Epub 2006 May 30. PMID 16781373
- [Background] Baron AD. Hemodynamic actions of insulin. Am J Physiol. 1994 Aug;267(2 Pt 1):E187-202. doi: 10.1152/ajpendo.1994.267.2.E187. PMID 8074198
- [Background] Baron AD, Laakso M, Brechtel G, Edelman SV. Mechanism of insulin resistance in insulin-dependent diabetes mellitus: a major role for reduced skeletal muscle blood flow. J Clin Endocrinol Metab. 1991 Sep;73(3):637-43. doi: 10.1210/jcem-73-3-637. PMID 1874938
- [Background] Laakso M, Edelman SV, Brechtel G, Baron AD. Decreased effect of insulin to stimulate skeletal muscle blood flow in obese man. A novel mechanism for insulin resistance. J Clin Invest. 1990 Jun;85(6):1844-52. doi: 10.1172/JCI114644. PMID 2189893
- [Background] Laakso M, Edelman SV, Brechtel G, Baron AD. Impaired insulin-mediated skeletal muscle blood flow in patients with NIDDM. Diabetes. 1992 Sep;41(9):1076-83. doi: 10.2337/diab.41.9.1076. PMID 1499861
- [Background] Vollenweider P, Tappy L, Randin D, Schneiter P, Jequier E, Nicod P, Scherrer U. Differential effects of hyperinsulinemia and carbohydrate metabolism on sympathetic nerve activity and muscle blood flow in humans. J Clin Invest. 1993 Jul;92(1):147-54. doi: 10.1172/JCI116542. PMID 8325979
- [Background] Raitakari M, Knuuti MJ, Ruotsalainen U, Laine H, Makea P, Teras M, Sipila H, Niskanen T, Raitakari OT, Iida H, Harkonen R, Wegelius U, Yki-Jarvinen H, Nuutila P, et al. Insulin increases blood volume in human skeletal muscle: studies using [15O]CO and positron emission tomography. Am J Physiol. 1995 Dec;269(6 Pt 1):E1000-5. doi: 10.1152/ajpendo.1995.269.6.E1000. PMID 8572189
- [Background] Raitakari M, Nuutila P, Knuuti J, Raitakari OT, Laine H, Ruotsalainen U, Kirvela O, Takala TO, Iida H, Yki-Jarvinen H. Effects of insulin on blood flow and volume in skeletal muscle of patients with IDDM: studies using [15O]H2O, [15O]CO, and positron emission tomography. Diabetes. 1997 Dec;46(12):2017-21. doi: 10.2337/diab.46.12.2017. PMID 9392489
- [Background] Tack CJ, Ong MK, Lutterman JA, Smits P. Insulin-induced vasodilatation and endothelial function in obesity/insulin resistance. Effects of troglitazone. Diabetologia. 1998 May;41(5):569-76. doi: 10.1007/s001250050948. PMID 9628275
- [Background] Yki-Jarvinen H, Utriainen T. Insulin-induced vasodilatation: physiology or pharmacology? Diabetologia. 1998 Apr;41(4):369-79. doi: 10.1007/s001250050919. No abstract available. PMID 9562340
- [Background] Taddei S, Virdis A, Mattei P, Natali A, Ferrannini E, Salvetti A. Effect of insulin on acetylcholine-induced vasodilation in normotensive subjects and patients with essential hypertension. Circulation. 1995 Nov 15;92(10):2911-8. doi: 10.1161/01.cir.92.10.2911. PMID 7586259
- [Background] Bonadonna RC, Saccomani MP, Del Prato S, Bonora E, DeFronzo RA, Cobelli C. Role of tissue-specific blood flow and tissue recruitment in insulin-mediated glucose uptake of human skeletal muscle. Circulation. 1998 Jul 21;98(3):234-41. doi: 10.1161/01.cir.98.3.234. PMID 9697823
- [Background] Steinberg HO, Brechtel G, Johnson A, Fineberg N, Baron AD. Insulin-mediated skeletal muscle vasodilation is nitric oxide dependent. A novel action of insulin to increase nitric oxide release. J Clin Invest. 1994 Sep;94(3):1172-9. doi: 10.1172/JCI117433. PMID 8083357
- [Background] Baron AD, Brechtel-Hook G, Johnson A, Cronin J, Leaming R, Steinberg HO. Effect of perfusion rate on the time course of insulin-mediated skeletal muscle glucose uptake. Am J Physiol. 1996 Dec;271(6 Pt 1):E1067-72. doi: 10.1152/ajpendo.1996.271.6.E1067. PMID 8997227
- [Background] Zhang L, Vincent MA, Richards SM, Clerk LH, Rattigan S, Clark MG, Barrett EJ. Insulin sensitivity of muscle capillary recruitment in vivo. Diabetes. 2004 Feb;53(2):447-53. doi: 10.2337/diabetes.53.2.447. PMID 14747297
- [Background] Eggleston EM, Jahn LA, Barrett EJ. Hyperinsulinemia rapidly increases human muscle microvascular perfusion but fails to increase muscle insulin clearance: evidence that a saturable process mediates muscle insulin uptake. Diabetes. 2007 Dec;56(12):2958-63. doi: 10.2337/db07-0670. Epub 2007 Aug 24. PMID 17720897
- [Background] Inyard AC, Clerk LH, Vincent MA, Barrett EJ. Contraction stimulates nitric oxide independent microvascular recruitment and increases muscle insulin uptake. Diabetes. 2007 Sep;56(9):2194-200. doi: 10.2337/db07-0020. Epub 2007 Jun 11. PMID 17563063
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Vincent MA, Barrett EJ, Lindner JR, Clark MG, Rattigan S. Inhibiting NOS blocks microvascular recruitment and blunts muscle glucose uptake in response to insulin. Am J Physiol Endocrinol Metab. 2003 Jul;285(1):E123-9. doi: 10.1152/ajpendo.00021.2003. PMID 12791603
- [Background] Clerk LH, Vincent MA, Barrett EJ, Lankford MF, Lindner JR. Skeletal muscle capillary responses to insulin are abnormal in late-stage diabetes and are restored by angiotensin-converting enzyme inhibition. Am J Physiol Endocrinol Metab. 2007 Dec;293(6):E1804-9. doi: 10.1152/ajpendo.00498.2007. Epub 2007 Oct 2. PMID 17911341
- [Background] Rattigan S, Clark MG, Barrett EJ. Acute vasoconstriction-induced insulin resistance in rat muscle in vivo. Diabetes. 1999 Mar;48(3):564-9. doi: 10.2337/diabetes.48.3.564. PMID 10078557
- [Background] Lauer T, Heiss C, Balzer J, Kehmeier E, Mangold S, Leyendecker T, Rottler J, Meyer C, Merx MW, Kelm M, Rassaf T. Age-dependent endothelial dysfunction is associated with failure to increase plasma nitrite in response to exercise. Basic Res Cardiol. 2008 May;103(3):291-7. doi: 10.1007/s00395-008-0714-3. Epub 2008 Mar 17. PMID 18347836
- [Background] Selvin E, Bolen S, Yeh HC, Wiley C, Wilson LM, Marinopoulos SS, Feldman L, Vassy J, Wilson R, Bass EB, Brancati FL. Cardiovascular outcomes in trials of oral diabetes medications: a systematic review. Arch Intern Med. 2008 Oct 27;168(19):2070-80. doi: 10.1001/archinte.168.19.2070. PMID 18955635
- [Background] Agarwal N, Rice SP, Bolusani H, Luzio SD, Dunseath G, Ludgate M, Rees DA. Metformin reduces arterial stiffness and improves endothelial function in young women with polycystic ovary syndrome: a randomized, placebo-controlled, crossover trial. J Clin Endocrinol Metab. 2010 Feb;95(2):722-30. doi: 10.1210/jc.2009-1985. Epub 2009 Dec 8. PMID 19996308
- [Background] Naka KK, Kalantaridou SN, Kravariti M, Bechlioulis A, Kazakos N, Calis KA, Makrigiannakis A, Katsouras CS, Chrousos GP, Tsatsoulis A, Michalis LK. Effect of the insulin sensitizers metformin and pioglitazone on endothelial function in young women with polycystic ovary syndrome: a prospective randomized study. Fertil Steril. 2011 Jan;95(1):203-9. doi: 10.1016/j.fertnstert.2010.06.058. Epub 2010 Aug 4. PMID 20684955
- [Background] Zou MH, Kirkpatrick SS, Davis BJ, Nelson JS, Wiles WG 4th, Schlattner U, Neumann D, Brownlee M, Freeman MB, Goldman MH. Activation of the AMP-activated protein kinase by the anti-diabetic drug metformin in vivo. Role of mitochondrial reactive nitrogen species. J Biol Chem. 2004 Oct 15;279(42):43940-51. doi: 10.1074/jbc.M404421200. Epub 2004 Jul 19. PMID 15265871 (Retraction: PMID 31492733 J Biol Chem. 2019 Sep 6;294(36):13525)
- [Background] Xie Z, Zhang J, Wu J, Viollet B, Zou MH. Upregulation of mitochondrial uncoupling protein-2 by the AMP-activated protein kinase in endothelial cells attenuates oxidative stress in diabetes. Diabetes. 2008 Dec;57(12):3222-30. doi: 10.2337/db08-0610. Epub 2008 Oct 3. PMID 18835932
- [Background] Katzmarzyk PT, Church TS, Blair SN. Cardiorespiratory fitness attenuates the effects of the metabolic syndrome on all-cause and cardiovascular disease mortality in men. Arch Intern Med. 2004 May 24;164(10):1092-7. doi: 10.1001/archinte.164.10.1092. PMID 15159266
- [Background] Allen JD, Geaghan JP, Greenway F, Welsch MA. Time course of improved flow-mediated dilation after short-term exercise training. Med Sci Sports Exerc. 2003 May;35(5):847-53. doi: 10.1249/01.MSS.0000064931.62916.8A. PMID 12750596
- [Background] Sugawara J, Otsuki T, Tanabe T, Hayashi K, Maeda S, Matsuda M. Physical activity duration, intensity, and arterial stiffening in postmenopausal women. Am J Hypertens. 2006 Oct;19(10):1032-6. doi: 10.1016/j.amjhyper.2006.03.008. PMID 17027823
- [Background] Miyaki A, Maeda S, Yoshizawa M, Misono M, Saito Y, Sasai H, Endo T, Nakata Y, Tanaka K, Ajisaka R. Effect of weight reduction with dietary intervention on arterial distensibility and endothelial function in obese men. Angiology. 2009 Jun-Jul;60(3):351-7. doi: 10.1177/0003319708325449. Epub 2008 Nov 19. PMID 19022788

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects failed the screening. 2 subjects voluntarily withdrew.
Groups:
- Placebo, Then Metformin: 12 weeks of Placebo tablet 3 x daily then 8 week washout then 12 weeks of metformin 500 mg 3x daily
- Metformin, Then Placebo: 12 weeks of metformin 500 mg tablet 3 x daily then 8 week washout then 12 weeks of placebo 3x daily
Period: Overall Study
Arm/Group | Placebo, Then Metformin | Metformin, Then Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, Then Metformin: 12 weeks of Placebo tablet 3 x daily, then a 8 week washout, then 12 weeks Metformin tablet 3 X daily
- Metformin, Then Placebo: 12 weeks of Metformin tablet 850 mg 3 x daily, then 8 week washout , then 12 weeks Placebo tablet 3X daily
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Metformin | Metformin, Then Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation - Endothelial Function
Description: brachial artery ultrasonography % flow-mediated dilatation (FMD) for assessing endothelial function before and after an insulin clamp to assess insulin's effect on the vasculature
Time Frame: before and after 12 weeks on placebo or metformin
Measure: Mean (Standard Error); unit: percentage of artery dilation
Groups:
- Pre and Post Placebo 12 Weeks: measured % dilation in response to shear stress before and after 2 hour insulin clamp which is performed before and after 12 weeks of Placebo tablets 3X daily
- Pre and Post Metformin 12 Weeks: measured % dilation in response to shear stress before and after 2 hour insulin clamp which is performed before and after 12 weeks of Metformin tablets 3X daily
Arm/Group | Pre and Post Placebo 12 Weeks | Pre and Post Metformin 12 Weeks
Number analyzed (Participants) | 11 | 11
percentage of artery dilation | 6.1 (1.1) | 6.2 (1.1)
Statistical Analysis 1: Comparison: Pre and Post Placebo 12 Weeks vs Pre and Post Metformin 12 Weeks; Test type: Equivalence — equivalence defined as less that 2 SD in FMD between 2 treatments; p > 0.05, t-test, 2 sided — FMD % change exceeded the threshold of our statistical significance test, i.e. the null hypothesis that there was no effect of metformin remained tenable

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Placebo | Metformin
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No